CLINICAL TRIAL: NCT03432767
Title: Investigating the Association of Shock Index and Hemoglobin Variation With Postpartum Hemorrhage After Vaginal Deliveries: A Prospective Cohort Study
Brief Title: Investigating the Association of Shock Index and Hemoglobin Variation With Postpartum Hemorrhage After Vaginal Deliveries
Status: Completed | Type: Observational
Sponsor: Samuel Lunenfeld Research Institute, Mount Sinai Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 18-03
Record Dates: First submitted 2018-02-05; First posted 2018-02-14 (Actual); Last update posted 2019-04-16 (Actual); Status verified 2019-04

CONDITIONS: Postpartum Hemorrhage
Keywords: pregnancy; postpartum hemorrhage; vaginal delivery; shock index; hemoglobin
MeSH Terms: conditions — Postpartum Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Women having a vaginal delivery: A non-invasive hemoglobin monitor will be attached to the patient's finger and kept on for 2 hours after she delivers. Heart rate and blood pressure will be measured every 10 minutes.
  Interventions: Device: Non-invasive hemoglobin monitor

INTERVENTIONS:
Device: Non-invasive hemoglobin monitor

SUMMARY:
Postpartum hemorrhage (PPH) is a leading cause of maternal mortality and morbidity, and is most commonly caused by poor uterine tone after delivery of the baby and placenta. Currently, a lack of early identification of PPH also results in delayed treatment, with an increase in morbidity. The investigators propose that 2 non-invasive methods may provide monitoring for early and accurate detection of PPH. These methods include shock index (SI) and continuous hemoglobin (Hb) monitoring. SI is defined as heart rate divided by systolic blood pressure, and can be used as a marker to predict the severity of hypovolemic shock. Continuous Hb monitoring can now be done using a non-invasive probe that is placed on the patient's finger. It provides real-time Hb values, rather than having to draw blood and wait for a lab test.

The investigators hypothesize that SI will have a stronger association with postpartum blood loss than Hb variation.

DETAILED DESCRIPTION:
The investigators believe that trends in patient-specific SI combined with continuous SpHb monitoring, will be useful to identify PPH and the immediate need for pharmacotherapy, as well as the need for transfusion in obstetric patients undergoing vaginal deliveries. The investigators expect shock index to increase and SpHb levels to decrease with increasing blood loss after delivery. The compensatory hemodynamic response may start early, however, Hb variation may be delayed unless the patient is transfused with crystalloids. Also autotransfusion after delivery may influence these measures. It is unknown which one of the two indicators, SI or SpHb, has a stronger association with blood loss after vaginal delivery.

It is already established that both SI and SpHb are independent, clinically useful markers indicating significant blood loss in elective cesarean delivery and trauma. This study would assess their utility in the recognition and management of obstetric hemorrhage following normal vaginal delivery, where early recognition and resuscitation reduces the risk of progressing to hemorrhagic shock, disseminated intravascular coagulation and death.

ELIGIBILITY:
Inclusion Criteria:

* patients who give written consent to participate in this study
* all term laboring patients including spontaneous and induced labor (gestational age >37 weeks) undergoing spontaneous vaginal delivery or instrumental delivery

Exclusion criteria

* patients who refuse to give written informed consent
* patients with cardiac rhythm abnormalities or cardiac diseases
* patients undergoing elective/emergency CD
* patients with jaundice
* patients with abnormal Hb-->Such as Sickle cell disease and Thalassemia
* patients with peripheral vascular disease
* patients with hypertension and preeclampsia
* patients on medications affecting blood pressure such as anti hypertensives (including Magnesium Sulphate), and those affecting HR (including beta blockers)

Ages: 16 Years to 50 Years | Sex: Female
Age Groups: Child, Adult
Study Population: Women having an expected vaginal delivery
Sampling Method: Non-Probability Sample
Enrollment: 67 (Actual)
Dates: Start 2016-02-16 (Actual); Primary Completion 2019-01-10 (Actual); Study Completion 2019-01-11 (Actual)

PRIMARY OUTCOMES:
Shock index values | 2 hours
  Calculated shock index (heart rate/systolic blood pressure) every 10 minutes from delivery until 2 hours postpartum.
Hemoglobin values | 2 hours
  Spectrophotometric hemoglobin values from a non-invasive monitor, recorded every 10 minutes from delivery until 2 hours postpartum.

SECONDARY OUTCOMES:
Estimated blood loss (calculated) | 24 hours
  Blood loss will be calculated through the difference in hematocrit values assessed prior to and at the end of 24 hours after the cesarean section.
Estimated blood loss (weight) | 2 hours
  Blood loss will be calculated by weighing the pads placed under the patient following delivery.
Administration of uterotonic medication | 24 hours
  Any oxytocin, ergonovine, carboprost, misoprostol administered following delivery
Blood transfusion | 24 hours
  The need for any transfusion of blood product following delivery.
Surgical interventions | 24 hours
  The need for manual placental removal, laceration/episiotomy repair, Bakri balloon, uterine artery ligation, hysterectomy, uterine artery/internal iliac artery embolization
ICU admission | 24 hours
  The need for admission to ICU following delivery

CONTACTS AND LOCATIONS:
Overall Officials: Mrinalini Balki, MD, Principal Investigator — MOUNT SINAI HOSPITAL
Locations (1):
- Mount Sinai Hospital, Toronto, Ontario, Canada

IPD SHARING:
Plan to Share IPD: No